CLINICAL TRIAL: NCT06530381
Title: Comparison of the Effects of Pilates Exercises Applied With Face-to-Face and Telerehabilitation Methods on Menstrual Pain
Brief Title: Effects of Pilates Exercises Applied With Face-to-Face and Telerehabilitation on Menstrual Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Duygu Şahin Altaç, PT, MSc., Halic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28.07.2024-MÜ
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Menstrual Pain
MeSH Terms: conditions — Dysmenorrhea | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Pilates Exercises Applied With Face-to-Face
  Interventions: Other: Pilates Exercises With Face-to-Face
- Group 2 (Experimental): Pilates Exercises Applied With Telerehabilitation
  Interventions: Other: Pilates Exercises With Telerehabilitation

INTERVENTIONS:
Other: Pilates Exercises With Face-to-Face — The exercise program includes a warm-up period; exercises performed in the supine position, bridge, side-lying position, prone position, quadripedal position and sitting positions, and a cool-down period. Exercises are performed face to face.
  Arms: Group 1
Other: Pilates Exercises With Telerehabilitation — The exercise program includes a warm-up period; exercises performed in the supine position, bridge, side-lying position, prone position, quadripedal position and sitting positions, and a cool-down period. Exercises are performed as telerehabilitation.
  Arms: Group 2

SUMMARY:
Pain is one of the most common symptoms of menstrual syndrome that significantly affects quality of life. The aim of our study is to compare the effect of Pilates on menstrual pain and the effectiveness of the applications within themselves.

DETAILED DESCRIPTION:
20 women experiencing severe pain during menstruation were randomized into two groups. The same exercise program is applied to 10 participants face-to-face, and to 10 participants via telerehabilitation. Exercises are applied for 6 weeks, 2 days a week. Visual Analog Scale (VAS) is used for pain assessment, SF-36 Short Form is used to assess quality of life, and Menstrual Attitude Scale is used to assess symptoms in the premenstrual/menstrual period. Evaluations are performed twice in total, before and after treatment. Statistical analysis will be performed with SPSS 24.0 program. If the data is parametric, paired sample t-test will be used for within-group evaluation; independent sample t-test will be used for between-group evaluation. If the data is non-parametric, Wilson test will be used for within-group evaluation and Mann Whitney U test will be used for between-group evaluation.

ELIGIBILITY:
Inclusion Criteria:

* People between the ages of 18-30 who have a continuing menstrual cycle.
* Women with menstrual pain VAS>5.
* People with regular menstrual cycles.

Exclusion Criteria:

* Being in menopause.
* Using birth control pills.
* Taking hormone therapy.
* Having exercise intolerance.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only women
Enrollment: 20 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | at baseline and at week 6.
  VAS is used for subjective assessment of pain. VAS scores are evaluated on a scale of 1-10. 1-3 indicates mild pain, 4-6 indicates moderate pain, 7-8 indicates severe pain, and 9-10 indicates very severe and unbearable pain.Individuals with VAS>5 are included in the study.
Short-Form 36 (SF-36) | at baseline and at week 6.
  The SF-36 scale is used for quality of life assessment. This scale basically includes 8 subject scales. Each subject title is scored between 0-100. The scale has positive scoring, as the score increases, the quality of life also increases.
Menstrual Attitude Scale (MAS) | at baseline and at week 6.
  MAS is used to evaluate symptoms in the premenstrual/menstrual period. MAS consists of 5 main topics and a total of 33 sub-items. MAS is a scale that includes both positive and negative items.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Şahin Altaç, PT, MSc., Principal Investigator — Halic University
Locations (1):
- Halic University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Unsal A, Ayranci U, Tozun M, Arslan G, Calik E. Prevalence of dysmenorrhea and its effect on quality of life among a group of female university students. Ups J Med Sci. 2010 May;115(2):138-45. doi: 10.3109/03009730903457218. PMID 20074018
- [Result] Daley A. The role of exercise in the treatment of menstrual disorders: the evidence. Br J Gen Pract. 2009 Apr;59(561):241-2. doi: 10.3399/bjgp09X420301. No abstract available. PMID 19341553
- [Result] Kirthika S V, S S, G MK, S R, Rnv D, P SS. Comparing Pilates and Gym Ball Exercises for Primary Dysmenorrhea Management: An Empirical Study. Cureus. 2024 Apr 28;16(4):e59184. doi: 10.7759/cureus.59184. eCollection 2024 Apr. PMID 38807793